CLINICAL TRIAL: NCT05304026
Title: Optimizing CO2 Injection Technique for Renal Artery Detection in Endovascular Abdominal Aortic Aneurysm Repair
Brief Title: Optimizing CO2 Injection Technique for EVAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Enrico Gallitto, Principal Investigator, University of Bologna
Other Study IDs: CO2 IT
Record Dates: First submitted 2022-03-03; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Abdominal Aortic Aneurysm; Endovascular Aortic Repair
Keywords: CO2; contrast medium; angiography
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Population: The group includes all patients undergoing EVAR, each patient is considered as both case and control of himself as the two CO2 injection techniques, through the 5F pigtail and through the 5F introducer, are both used during the procedure.
  Interventions: Device: Technique 1; Device: Technique 2; Device: Technique 3; Device: Technique 4

INTERVENTIONS:
Device: Technique 1 — It refers to CO2 digital subtraction angiographies performed at the beginning of the procedure through a 5F pigtail catheter placed at the level of renal arteries to identify the lowest renal artery.
Device: Technique 2 — It refers to CO2 digital subtraction angiographies performed at the beginning of the procedure through a 5F introducer placed at the end of the proximal sealing zone to identify the lowest renal artery.
Device: Technique 3 — It refers to CO2 digital subtraction angiographies performed at the end of the procedure through a 5F pigtail catheter through the pigtail catheter placed at the level of renal arteries.
Device: Technique 4 — It refers to CO2 digital subtraction angiographies performed at the end of the procedure through a 5F introducer placed at the level of the contralateral iliac limb.

SUMMARY:
Automated carbon dioxide (CO2) angiography is considered a safe diagnostic alternative to standard iodinated contrast medium (ICM) for endovascular aortic repair (EVAR) of abdominal aortic aneurysm (AAA), especially in patients with preoperative renal function impairment.

Recent literature experiences describe the use of automated CO2 angiography in EVAR.

One of the main issues of CO2 angiography is the inability to detect the origin of the lowest renal artery (proximal neck visualization) that was estimated up to 38%.

In these experiences, the CO2 automated angiography is usually performed by a 5F pigtail catheter placed at renal arteries level.

The aim of the study is to evaluate the efficacy of a new automated CO2 injection technique by a 5F introducer (single hole catheter) positioned at the distal level of the proximal neck in detecting both renal arteries in the first diagnostic and completion angiographies.

DETAILED DESCRIPTION:
Endovascular aneurysm repair is currently a wide spread therapeutic option due to a lower 30-day morbidity/mortality compared with open repair (OR), especially in patients with high surgical risk. The routinary EVAR technique requires the use of iodinated contrast medium (ICM) which can cause contrast induced-acute kidney injure (CI-AKI). The incidence of CI-AKI after EVAR is estimated between 2% and 16% although renal insult can also be caused by microembolization, unplanned renal (or polar) artery coverage, renal artery lesion (as dissection) or post-operative inflammatory reaction.

In the past few years, several studies pointed out the importance of reducing the amount of iodinated contrast medium injected and proposed carbon dioxide (CO2) as an alternative to partially or completely replace ICM, especially in patients with preoperative chronic renal impairment.

According with the literature, manual or automatic CO2 injection provides a good quality imaging of both proximal and distal sealing zone in standard EVAR procedures and, combined with fusion imaging, allows to perform juxta and pararenal abdominal aortic aneurysm repair with fenestrated endograft reducing the total amount of ICM required to the procedure.

The most relevant limit to the use of CO2 is the inability to identify the proximal landing zone and the lowest renal artery that occurs in a significant number of cases (38.7%).

This limit could be related to the physical property of CO2 because, differently from ICM, it is a gas that does not completely fill the aortic lumen but it floats in the anterior portion of the aneurysmatic sac and does not allow the detection of renal arteries with a posterior origin.

The automated CO2 injection is commonly performed using a pigtail catheter (5F/65mm length) placed at the renal arteries level.

The primary end point of the study is to identify an alternative and effective method of CO2 injection, using an automatic system through the digital Angiodroid injection system (Angiodroid Srl, San Lazzaro, Bologna) connected to a 5F introducer placed at the distal portion of infra-renal neck that allows the identification of the lowest renal artery.

This is a prospective, single center, observational, case-control study, in which each patient is the control of himself because during the procedure 2 angiographic CO2 techniques (angiography by pig tail vs 5 F introducer) are performed and compared.

All patients underwent a preoperative computed tomography angiography (CTA) within 3 months before the procedure. The images are analyzed using a dedicated software for vessel analysis (3Mensio TM, Vascular Imaging Bilthover, Netherlands) and the AAA volume is calculated using the same software by selecting points of the external aortic wall and internal aortic lumen from the lower renal artery to the aortic bifurcation.

The level of renal arteries and aortic bifurcation are evaluated on preoperative CTA reconstructions and matched with vertebral bone landmarks.

At the beginning of the procedure two CO2 DSA will be performed: the first one through the pigtail placed at the level of renal arteries and the second one through a 5F introducer placed at the end of the proximal sealing zone in order to identify the lowest renal artery and compare the quality of the images obtained.

The same way, at the end of the procedure after the endograft deployment, two CO2 DSA will be performed: the first one through the pigtail catheter placed at the level of renal arteries and the second one through the 5F introducer placed at the level of the contralateral iliac limb.

The investigators prospectively collect clinical and morphological preoperative, intraoperative and postoperative data as shown in the table above.

Clinical characteristics: age years, sex, hypertension (systolic blood pressure ≥140 or/and diastolic ≥90 mmHg, or specific therapy), dyslipidemia (total cholesterol ≥200 mg/dl or low density lipoprotein ≥120 mg/dl or specific therapy), diabetes mellitus (pre-diagnosed in therapy with oral hypoglycemic drugs or with insulin), current smoking, coronary artery disease (defined as a history of angina pectoris, myocardial infarction or coronary revascularization), chronic obstructive pulmonary disease (defined as chronic bronchitis or emphysema), chronic kidney disease (glomerular filtration rate <60 ml/min), dialysis, pre and post-operative creatinine serum, ASA (American Society Anesthesiologic classification), medical therapy (antiplatelet types, anticoagulant therapy, statin therapy, anti-hypertensive medical therapy).

Morphological characteristics: aneurysm diameter, aneurysm volume, aneurysm neck features according to Chaickof classification, iliac axes features according to Chaickof classification, renal arteries number and clock position, hypogastric arteries patency, aortic carrefour diameter.

Intraoperative data: anesthesia (general or spinal), vascular access (surgical or percutaneous), endograft features (bi- or tri-modular, suprarenal fixation, proximal diameter of the endograft, left and right iliac limb diameter, embolization of the aneurysmatic sac, coils number, hypogastric embolization or coverage, other adjunctive maneuvers as iliac axes stenting), type and amount of contrast medium, fluoroscopy time, dose area product (DAP) (fluoroscopy DAP, DSA DAP and total DAP), renal arteries detection at the beginning of the procedure with CO2 DSA from 5F pigtail and 5F introducer, renal and hypogastric arteries and endoleaks detection at the end of the procedure with CO2 DSA from 5F pigtail and 5F introducer (as explained before).

Post-operative data: complications related to CO2 injection rate (nausea, vomit, abdominal pain, hypotension), endoleaks at the discharge, perioperative mortality, 30-days mortality, 30-days medical or surgical complications, 30-days reintervention rate, 30-days renal function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with asymptomatic infrarenal abdominal aortic aneurysm admitted to the S. Orsola - Malpighi Hospital for a planned EVAR procedure. All patients underwent a preoperative computed tomography angiography (CTA) with a <2mm slices.

Exclusion Criteria:

* Patients with contraindication for CO2 (cardiac septal defects, pulmonary arteriovenous malformations, pulmonary hypertension, severe emphysema)
* Patients requiring advanced aortic repair (FEVAR, BEVAR)
* Urgent cases

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All elective patients with asymptomatic infrarenal abdominal aortic aneurysm (according to the ESVS guidelines) undergoing EVAR with automated CO2 digital subtraction angiography (DSA) from January 2021.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Aortic neck detection | At the moment of CO2 injection during the procedure
  Define the efficacy of the alternative CO2 injection technique in the detection of renal arteries in those cases when the usual technique doesn't succeed.
Procedure success | At the moment of CO2 injection during the procedure
  Define the efficacy of the alternative CO2 injection technique in the detection of renal arteries, hypogastric arteries and endoleaks at the final angiography in those cases when the usual technique doesn't succeed.

SECONDARY OUTCOMES:
CO2 complications | within 30 days from the procedure
  Evaluate CO2 induced complications rate
Mortality | within 30 days from the procedure
  Evaluate 30-day mortality related to procedure
Adverse events | within 30 days from the procedure
  Assessment of any cardiopulmonary and renal events related to the procedure
Rate of early reintervention | within 30 days from the procedure
  Any re-intervention needed after the procedure and the specific reason

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Gallitto, MD, PhD, Principal Investigator — University of Bologna
Locations (1):
- University of Bologna, Bologna, Emilia-Romagna, Italy

REFERENCES:
- [Background] Mascoli C, Faggioli G, Gallitto E, Vento V, Pini R, Vacirca A, Indelicato G, Gargiulo M, Stella A. Standardization of a Carbon Dioxide Automated System for Endovascular Aortic Aneurysm Repair. Ann Vasc Surg. 2018 Aug;51:160-169. doi: 10.1016/j.avsg.2018.01.099. Epub 2018 Mar 6. PMID 29522871
- [Background] Gallitto E, Faggioli G, Vacirca A, Pini R, Mascoli C, Fenelli C, Logiacco A, Abualhin M, Gargiulo M. The benefit of combined carbon dioxide automated angiography and fusion imaging in preserving perioperative renal function in fenestrated endografting. J Vasc Surg. 2020 Dec;72(6):1906-1916. doi: 10.1016/j.jvs.2020.02.051. Epub 2020 Apr 8. PMID 32276017
- [Background] Mascoli C, Faggioli G, Gallitto E, Vento V, Indelicato G, Pini R, Vacirca A, Stella A, Gargiulo M. The Assessment of Carbon Dioxide Automated Angiography in Type II Endoleaks Detection: Comparison with Contrast-Enhanced Ultrasound. Contrast Media Mol Imaging. 2018 Mar 26;2018:7647165. doi: 10.1155/2018/7647165. eCollection 2018. PMID 29780288
- [Background] Vacirca A, Faggioli G, Mascoli C, Gallitto E, Pini R, Spath P, Logiacco A, Palermo S, Gargiulo M. CO2 Automated Angiography in Endovascular Aortic Repair Preserves Renal Function to a Greater Extent Compared with Iodinated Contrast Medium. Analysis of Technical and Anatomical Details. Ann Vasc Surg. 2022 Apr;81:79-88. doi: 10.1016/j.avsg.2021.10.039. Epub 2021 Nov 14. PMID 34785338